CLINICAL TRIAL: NCT07005401
Title: What Determines the Feasibility and Surgical Margin Quality of Sublobar Resection for Small-sized Non-small Cell Lung Cancer?
Brief Title: Factors Determine the Feasibility and Surgical Margin Quality of Sublobar Resection for Non-small Cell Lung Cancer?
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Liang Chen, Professor, The First Affiliated Hospital with Nanjing Medical University
Other Study IDs: TSCI 002
Record Dates: First submitted 2025-05-27; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-small cell lung cancer; Segmentectomy; Wedge resection; Margin quality
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients undergoing eligible sublobar resection: A surgical margin ≥ the maximum tumor diameter was considered sufficient. Sublobar resection with a sufficient surgical margin was considered eligible.
- Patients undergoing lobectomy or ineligible sublobar resection: Patients who underwent lobectomy or received ineligible sublobar resection (sublobar resection with an insufficient surgical margin: less than the maximum tumor diameter)

SUMMARY:
Sublobar resection (SR) has been recognized as non-inferior to lobectomy for small-sized non-small cell lung cancer (NSCLC). This study aimed to systematically identify the potential factors influencing the feasibility and surgical margin quality of SR for small-sized NSCLC.

Patients with small-sized NSCLC (≤2 cm) who underwent SR or lobectomy between 2020 and 2023 were screened. Surgical procedures were determined by discussion under the guidance of 3D-CTBA. A surgical margin ≥ the maximum tumor diameter was considered sufficient. SR with a sufficient surgical margin was considered eligible. Univariate and multivariate logistic regression analyses were performed to identify factors affecting the feasibility and margin quality of SR.

DETAILED DESCRIPTION:
Patients with small-sized pulmonary nodules who underwent lobectomy or SR between 2020 and 2023 in a single surgical team were retrospectively screened. All the surgical approach was jointly determined by three experienced surgeons (at least 15 years, Doctor Liang Chen, Weibing Wu and Zhicheng He). Patients satisfied with the following criteria were initially reserved: (1) the maximum nodule diameter ≤ 2 cm; (2) single malignant nodule; (3) intentional resection; (4) histopathological confirmed primary NSCLC. Further, patients with (1) interlobar lesions; (2) nodules in the right middle lobe; (3) receiving neoadjuvant before surgery; (4) poor CT quality were excluded.

ELIGIBILITY:
Inclusion Criteria:

* the maximum nodule diameter ≤ 2 cm
* single malignant nodule
* intentional resection
* histopathological confirmed primary non-small cell lung cancer

Exclusion Criteria:

* interlobar lesions
* nodules located in the right middle lobe
* receiving neoadjuvant before surgery
* poor CT quality were excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with small-sized pulmonary nodules who underwent lobectomy or sublobar resection between 2020 and 2023 in a single surgical team were retrospectively screened.
Sampling Method: Non-Probability Sample
Enrollment: 1064 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
surgical margin quality | Perioperative
  A surgical margin ≥ the maximum tumor diameter was considered sufficient.

CONTACTS AND LOCATIONS:
Overall Officials: Liang Chen, MD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No